CLINICAL TRIAL: NCT05279391
Title: Combined Administration of Inhaled DNase, Baricitinib and Tocilizumab as Rescue Treatment in Severe COVID-19 Patients
Brief Title: Combination of Inhaled DNase, Baricitinib and Tocilizumab in Severe COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Konstantinos Ritis, Professor of Internal Medicine, First Department of Internal Medicine, Democritus University of Thrace
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 87/08-04-2020; 16210/20-04-2021 (Other: University Hospital of Alexandroupolis, Greece)
Record Dates: First submitted 2022-03-11; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Severe Respiratory Failure
Keywords: COVID-19; Respiratory failure; Inhaled DNase; Baricitinib; Tocilizumab; Low molecular weight heparin; Dexamethasone; Anakinra
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Dexamethasone; Heparin, Low-Molecular-Weight; Interleukin 1 Receptor Antagonist Protein; tocilizumab; baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SOC (Active Comparator): Patients included in this arm treated with the standard of care (SOC), including dexamethasone plus heparin, with or without the addition of antibiotics and remdesivir
  Interventions: Drug: Dexamethasone; Drug: Low molecular weight heparin
- TOCI (Active Comparator): Patients included in this arm treated with the SOC plus Tocilizumab (single IV dose: 8mg/kg)
  Interventions: Drug: Dexamethasone; Drug: Low molecular weight heparin; Drug: Tocilizumab
- ANA (Active Comparator): Patients included in this arm treated with the SOC plus Anakinra (200mg twice daily IV for 3-6 days, then 100 mg/twice daily, for up to 10 days in total)
  Interventions: Drug: Dexamethasone; Drug: Low molecular weight heparin; Drug: Anakinra 100Mg/0.67Ml Inj Syringe
- COMBI (Active Comparator): Patients included in this arm treated with the SOC plus the combination of Tocilizumab, Baricitinib and inhaled DNase (COMBI) as a rescue treatment.
  Interventions: Drug: Dexamethasone; Drug: Low molecular weight heparin; Drug: Tocilizumab; Drug: Baricitinib; Drug: Dornase Alfa Inhalant Product

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 6-8 mg once daily
Drug: Low molecular weight heparin — Therapeutic doses of LMWH (e.g. Tinzaparin 175IU/kg)
Drug: Anakinra 100Mg/0.67Ml Inj Syringe — IV administration of Anakinra 200 mg/twice daily for 3-6 days, then 100 mg/twice daily, for up to 10 days in total.
  Arms: ANA
Drug: Tocilizumab — IV administration of Tocilizumab as a single dose of 8mg/kg
  Arms: COMBI; TOCI
Drug: Baricitinib — 4 mg per os once daily, for up to 14 days (2 mg if GFR: 30 to <60 ml/min/1.73 m2)
  Arms: COMBI
Drug: Dornase Alfa Inhalant Product — Inh. 2,500 U/twice daily, for up to 14 days.
  Arms: COMBI

SUMMARY:
In patients with COVID-19, severe hypoxemic respiratory failure (SRF) leading to invasive mechanical ventilation (IMV), raises the mortality rate substantially. Thus, the management of patients with SRF to avoid intubation and intensive care admission is a challenging and crucial issue.

This study describes, as rescue/compassionate treatment, a therapeutic protocol based on the multi-mechanistic nature of severe COVID-19, using the combination of inhaled DNase, Baricitinib and Tocilizumab on top of standard of care (SOC) consisting of heparin and dexamethasone. COVID-19 patients with SRF who were treated with SOC, SOC plus Anakinra (ANA), and SOC plus Tocilizumab (TOCI) will be studied as comparators. Primary endpoint will be the reduction of the in-hospital mortality rate, whereas secondary endpoints concern intubation rate, days of hospitalization and overall survival as derived from the last follow-up visit, either in-office or remote.

This is a non-randomized, open-label, study, conducted in the First Department of Internal Medicine, University Hospital of Alexandroupolis, Greece.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients ≥18 years old, of any gender
2. positive polymerase-chain-reaction (PCR) test for SARS-CoV-2 RNA in nasopharyngeal swab
3. pulmonary infiltrates suggestive of COVID-19
4. severe respiratory failure (SRF) as defined by PaO2/FiO2<100 mm Hg
5. written informed consent from the patients or legal representatives for the current compassionate therapeutic protocol.

Exclusion Criteria:

1. need for intubation/IMV during the first 24 hours after the initiation of treatment
2. multi-organ failure,
3. systemic co-infection
4. SRF due to cardiac failure or fluid overload
5. glomerular filtration rate (GFR) <30 ml/min/1.73 m2)
6. any stage IV solid tumor or immunosuppression due to hematological disorders
7. any immunosuppressive therapy and/or chemotherapy during the last 30 days
8. low patient's functional performance as defined by a Palliative Performance Scale (PPS) score ≤30%
9. pregnancy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality rate | Through study completion, an average of 1 year
  To investigate whether the combined administration of inhaled DNase, Baricitinib and Tocilizumab, as a rescue treatment, reduces the in-hospital mortality rate in COVID-19 patients with severe respiratory failure compared to standard of care and other immunomodulatory treatments.

SECONDARY OUTCOMES:
Intubation rate | Through study completion, an average of 1 year
  To investigate whether the combined administration of inhaled DNase, Baricitinib and Tocilizumab, as a rescue treatment, reduces the intubation rate in COVID-19 patients with severe respiratory failure compared to standard of care and other immunomodulatory treatments.
Days of hospitalization | Through study completion, an average of 1 year
  To investigate whether the combined administration of inhaled DNase, Baricitinib and Tocilizumab, as a rescue treatment, reduces the days of hospitalization in COVID-19 patients with severe respiratory failure compared to standard of care and other immunomodulatory treatments.
Overall mortality rate | Follow-up (max: 52 weeks)
  To investigate whether the combined administration of inhaled DNase, Baricitinib and Tocilizumab, as a rescue treatment, affects overall survival in a follow up of a maximum 52 weeks in COVID-19 patients with severe respiratory failure compared to standard of care and other immunomodulatory treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece